CLINICAL TRIAL: NCT05819554
Title: Evaluation of Expression of Somatostatin Receptors and GH Receptor on Bone of Acromegalic Patients (ACRO-BONE)
Brief Title: Evaluation of Somatostatin Receptors and GH Receptor Expression on Bone of Acromegalic Patients (ACRO-BONE)
Acronym: ACRO-BONE
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5367
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-03

CONDITIONS: Evaluation of the Expression of Somatostatin Receptors and GH Receptor on Bone of Acromegalic Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Acromegaly patients
  Interventions: Procedure: Trans-sphenoidal surgery
- Non-secreting pituitary tumors affected patients
  Interventions: Procedure: Trans-sphenoidal surgery
- Secreting pituitary tumors affected patients
  Interventions: Procedure: Trans-sphenoidal surgery
- Healthy patients
  Interventions: Procedure: Trans-sphenoidal surgery

INTERVENTIONS:
Procedure: Trans-sphenoidal surgery — Surgical removal of pituitary tumor by trans-sphenoidal approach

SUMMARY:
Skeletal fragility is a frequent complication in patients with acromegaly. About 30% of patients with acromegaly can develop spontaneous vertebral fractures. Preliminary data show that patients suffering from acromegaly and treated with second generation somatostatin analogues (Pasireotide Lar) are more protected from the risk of vertebral fractures, compared to patients treated with other therapeutic lines (such as first generation analogues) . The molecular basis of this therapeutic effect on bone metabolism has not been identified. Since second generation somatostatin analogues preferentially bind somatostatin receptor subtype 5, while first generation analogues bind both subtypes 2 and 5, our work aims to evaluate the expression pattern of somatostatin receptors somatostatin on bone tissue of patients with acromegaly, comparing it with the bone receptor profile of a control group, composed of patients with non-secreting pituitary adenomas and prolactin and ACTH-secreting pituitary adenomas and healthy subjects undergoing septoplasty for nasal septum deviation .

ELIGIBILITY:
Inclusion Criteria:

* patients with pituitary adenoma, with indication for neurosurgical removal, in accordance with current guidelines;
* patients indicated for septoplasty, in accordance with current guidelines;
* availability of bone tissue, removed as per current clinical practice, during trans-nasosphenoidal surgery, for the molecular procedures required in the protocol
* patients older than 18 years.
* signature of the informed consent

Exclusion Criteria:

* patients suffering from bone pathologies, such as dysplastic syndromes, primary and secondary bone tumors.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will consist of 20 cases of patients with acromegaly and a control group consisting of 20 patients with non-secreting pituitary adenomas, 20 patients with secretory pituitary adenomas (10 cases of prolactinoma and 10 cases of Cushing's disease). and 20 healthy subjects (patients undergoing septoplasty for deviation of the nasal septum).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the expression pattern of somatostatin receptors on bone tissue of patients with acromegaly | 12 months

SECONDARY OUTCOMES:
Evaluation of the differences in the expression of SSTR2A between the group of acromegalic patients compared to the control group | 12 months
Evaluation of the differences in the expression of SSTR5 between the group of acromegalic patients compared to the control group | 12 months
Evaluation of the differences in the expression of the GH receptor between the group of acromegalic patients and the control group | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinnico Gemelli IRCCS, Roma, Italy